CLINICAL TRIAL: NCT05215158
Title: A Comparative Study of Intravenous Versus Peribulbar Administration of Dexmedetomidine for Strabismus Surgery in Adults
Brief Title: Intravenous Versus Peribulbar Dexmedetomidine for Strabismus Surgery in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 520/3/21
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Squint
MeSH Terms: conditions — Strabismus | interventions — Dexmedetomidine; Adrenergic alpha-2 Receptor Agonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peribulbar dexmedetomidine (Active Comparator): The peribulbar block will be done using a mixture of 4 ml Lidocaine 2%, 4 ml Bupivacaine 0.5%, and 2 ml normal saline containing 50 μg dexmedetomidine perineurally (30 patients).
  Interventions: Drug: Dexmedetomidine
- Intravenous dexmedetomidine (Active Comparator): The peribulbar block will be done using a mixture of 4 ml Lidocaine 2%, 4 ml Bupivacaine 0.5%, and 2 ml normal saline. Patients received 50 μg dexmedetomidine in 50 mL of normal saline administered as an infusion over 10 minutes, and given 10 minutes before the peribulbar block (30 patients).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — to compare perineural (peribulbar) dexmedetomidine versus intravenous (I.V.) dexmedetomidine when used as an adjuvant with local anesthesia in adult strabismus surgery.
  Other Names: alpha-2 agonist

SUMMARY:
Using various adjuvants has become a trend in regional anesthesia practice to improve the quality of anesthesia and prolong postoperative analgesia. Dexmedetomidine, an alpha-2 agonist has been proposed as a safe and effective adjunct capable of extending the duration of the single-shot block

DETAILED DESCRIPTION:
Strabismus (misalignment of the eye) results from a difference in extraocular muscle function. Consequently, two different images, one from each eye, are transmitted to the brain, resulting in a loss of visual depth. In adults, cosmetic appearance is the main issue but sudden occurrence of strabismus may cause diplopia because the brain cannot suppress the overlapping images. The goal of strabismus surgery is to align the eyes, reduce diplopia, and restore binocular vision Ophthalmic regional block can be used as the primary anesthetic technique for strabismus surgery. The advantages of ophthalmic regional blockade include a reduced incidence of oculocardiac reflex (OCR) and emergence agitation, postoperative analgesia, and decreased postoperative nausea and vomiting (PONV).

Using various adjuvants has become a trend in regional anesthesia practice to improve the quality of anesthesia and prolong postoperative analgesia. Dexmedetomidine, an alpha-2 agonist has been proposed as a safe and effective adjunct capable of extending the duration of the single-shot block.

Perineural dexmedetomidine, when added to bupivacaine, has been shown to potentiate its effects, providing a better quality of anesthesia and postoperative analgesia. Intravenous (I.V.) dexmedetomidine, when used during regional anesthesia, has been shown to prolong sensory and motor blockade in addition to sedation and postoperative analgesia.

No previous studies where different routes of dexmedetomidine have been compared in adult strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient planned to perform a unilateral strabismus surgery
2. Age: 20-60 years
3. American Society of Anesthesiologists class I and II

Exclusion Criteria:

1. patients under the age of 20
2. uncooperative patients
3. Patients with coagulopathy
4. patients who disincline to participate in the study will be excluded from the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | 12 hours
  The time gap between the abolition of the sensation using gauze soaked in cooled normal saline, or corneal reflex, and the first postoperative demand for analgesia

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aswan University Hospital, Aswān
  - Huda Fahmy, Aswān

REFERENCES:
- [Derived] Ghazaly HF, Hassan IE, Gabr AF, Dardeer TT, Alazhary MA. Intravenous Versus Peribulbar Dexmedetomidine as an Adjunct to Local Anesthetics in Strabismus Surgery: A Randomized, Double-blinded Clinical Trial. Pain Physician. 2024 Nov;27(8):E819-E827. PMID 39621979